CLINICAL TRIAL: NCT06230237
Title: Telephone Support vs. Self-guidance in an Internet-based Self-administered Psychological Program for the Treatment of Depression
Brief Title: Telephone Support vs. Self-guidance in an Internet-based Self-administered Psychological Program to Address Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitat Jaume I (Other)
Collaborators: Hospital Francesc de Borja (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FISABIO
Record Dates: First submitted 2022-04-19; First posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Depression
Keywords: Depression; Internet Based Intervention; Psychological Intervention; Professional Support; Mental Health; Self-guided
MeSH Terms: conditions — Depression; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Professional support (Active Comparator): Participants randomly assigned to this groups will receive the self-administered psychotherapy via the Internet a with telephone psychotherapeutic support.
  Interventions: Behavioral: Smiling is fun + professional support
- Non professional support (Active Comparator): Participants randomly assigned to this group will receive the self-administered psychotherapy via the Internet without telephone psychotherapeutic support.
  Interventions: Behavioral: Smiling is fun

INTERVENTIONS:
Behavioral: Smiling is fun + professional support — Participants will receive an intervention called Smiling is Fun; a cognitve-conductual online program with the most effective psychological procedures for depression and other techniques to promote coping ability, emotional regulation and resilience along 8 modules.
  While they do the online program, they will receive periodically professional support. The professional support will be contacts of 20 minutes long, will take place every two weeks and will last 3 months.
  Arms: Professional support
Behavioral: Smiling is fun — Participants will receive an intervention called Smiling is Fun; a cognitve-conductual online program with the most effective psychological procedures for depression and other techniques to promote coping ability, emotional regulation and resilience along 8 modules.
  Arms: Non professional support

SUMMARY:
Depression is a first level problem that poses a challenge for Primary Care (PC). The overload of care in this area requires lower-cost and more accessible alternatives. Internet-based self-applied cognitive behavioral treatments (CBCT) have demonstrated their efficacy and added advantages. The "Smiling is fun" program has been validated in Spanish PC and has demonstrated its usefulness and cost-effectiveness. Previous studies have shown that professional support or guidance increases the results of the TCCI.

The aim of the present study is to contrast, by means of a randomized controlled trial, aims to examine the effectiveness, adherence rates, and implementation process of Smiling is Fun to address depression in a PC setting considering the influence of telephone support vs no support.

Ultimately, the results of the study could help in the uptake of sustainable resources so that the population could gain better access to psychological interventions in mental health services.

DETAILED DESCRIPTION:
Background: Depression is already the leading psychological disability around the world, impairing daily life, well-being, and social functioning and leading to personal and social costs. Despite the effectiveness of Evidence-Based Psychological Practices (EBPP), a significant percentage of depressive individuals remain untreated, especially in Primary Care (PC) settings in Spain. There are numerous barriers that limit access to EBPPs, including high costs, professional training, and adherence problems. Information and Communication Technologies (ICTs) offer a cost-effective way to disseminate and scale EBPPs to address these barriers. The iCBT program Smiling is Fun has been demonstrated to be a cost-effective treatment for depression in various Randomized Control Trials. However, adherence and implementation problems in real-world settings need to be addressed. Implementation research can help evaluate these challenges by identifying facilitators and barriers to the implementation process in PC. In this regard, guided support has been pointed out as a possible key factor in addressing the population's mental health needs and promoting treatment adherence. Objective: The current study aims to examine the effectiveness, adherence rates, and implementation process of Smiling is Fun to address depression in a PC setting considering the influence of telephone support vs no support. Methods: The proposed research is a Hybrid Effectiveness-Implementation Type I study, with a two-armed randomized controlled design, which will test a clinical intervention for major depressive disorder while gathering information on its implementation in a real-world setting. The study will include adult patients with mild to moderate symptoms of depression. Participants will be randomly assigned to one of two groups: self-applied psychotherapy or self-applied psychotherapy with psychotherapeutic telephone support. The trial will recruit 100 patient participants, with a loss-to-follow-up rate of 30%. Discussion: A study protocol for a hybrid effectiveness-implementation study is presented with the aim to assess the implementation of Smiling is Fun for the treatment of depression in PC. The study evaluates the influence of telephone support during a self-administered intervention compared to unguided self-administration. The main goal is to address the barriers and facilitators of the implementation process and to promote treatment adherence. Ultimately, the results of the study could help in the uptake of sustainable resources so that the population could gain better access to psychological interventions in mental health services.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65 years.
* Ability to understand and read Spanish.
* Meet diagnostic criteria for major depressive disorder (DSM-5).
* Mild or moderate symptoms of the Spanish version of the Beck Depression Inventory-II (BDI-II) (14-19: mild depression; 20-28: moderate depression).
* Episode duration of more than two weeks.
* Have internet access at home and an email account.
* The diagnosis of major depressive disorder will be confirmed by the standardized MINI International Neuropsychiatric Interview.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Treatment efficacy | Pre-intervention, immediately after the intervention and follow-up (3,6 and 12 months).
  Change of depression symtpmatology through the Beck Depression Inventory (BDI-II).

SECONDARY OUTCOMES:
Quality of life related to health | Pre-intervention, immediately after the intervention and follow-up (3,6 and 12 months).
  The qualitiy of life related to health apsects will be measured using : EuroQol (EQ-5D) and Short Form Health Survey (SF-12)

OTHER OUTCOMES:
Adherence to the treatment | Immediately after the intervention
  The adherence to the treatment will be assessed according to the moduls done by the patient in the plataform
Implementation outcome: Feasibility | Immediately after the intervention
  Professionals' assessment: Feasibility of Intervention Measure (FIM) (Weiner et al., 2017). A four items scale on a 5-point Likert scale assess the feasibility of an intervention in a specific context. The FIM showed high levels of internal consistency (α =0,89) and test-retest reliability coefficients (α =0,88).
Implementation outcome: Acceptability | Immediately after the intervention
  Professionals' assessment: Acceptability of Intervention Measure (AIM) (Weiner et al., 2017). A 4-item scale (from 1= completely disagree to 5= completely agree) that assesses the perception of the stakeholders about the agreeableness of treatment in a specific context. The construct has shown good psychometric properties with high levels of internal consistency (α =0.89) and test-retest reliability (α =0.83).
Implementation outcome: Appropiateness | Immediately after the intervention
  Professionals' assessment: Intervention Appropriateness Measure (IAM) (Weiner et al., 2017). A 4-item scale (from 1= completely disagree to 5= completely agree) that measures the appropriateness of the intervention. The scale has shown good psychometric properties with high levels of internal consistency (α =0.87) and test-retest reliability (α =0.87)
Implementation outcome: Normalization | Immediately after the intervention
  Professionals' assessment: Normalization MeAsure Development Questionnaire (NoMAD) (Finch et al., 2018). Based on the Normalization Process Theory, the NoMAD, a questionnaire of 13 items 5-Likert scale (from strongly agree to strongly disagree), has been developed to assess the process of normalization (May et al., 2009). The NoMAD focuses on four dimensions: coherence, cognitive participation, collective action, and reflexive monitoring. This questionnaire has demonstrated high levels of internal consistency along the four dimensions (20 items) (alpha=0.89).
Implementation outcome: Attitudes Towards Psychological Online Intervention | Immediately after the intervention
  Professionals' assessment: Attitudes towards Psychological Online Interventions (APOI) (Schröder et al., 2015). A 16-item questionnaire, with a 5-point Likert scale, assesses attitudes toward IBT. The APOI explores four dimensions; "Skepticism and Perception of Risks", "Confidence in Effectiveness", "Technologization Threat" and "Anonymity Benefits". The scale has shown acceptable to good internal consistency (α=0.77) (Schröder et al., 2015).
Implementation outcome: Sustainability | Immediately after the intervention
  Professionals' assessment: Barriers and facilitators of the implementation (FBI). The FBI is a questionnaire specifically developed for this study and the study conducted by Lorente-Català et al. (2022). The questionnaire was created following the systematic review on EBT implementation barriers and facilitators among third sector organizations (Bach-Mortensen et al., 2018). As a result, 28 items assess the possible barriers, and 15 items evaluate the facilitators.
Implementation outcome: Satisfactions | Immediately after the intervention
  Client Satisfaction Questionnaire adapted to Internet-Based Interventions (CSQ-I; Boß et al., 2016). This 9-item questionnaire assesses participants' satisfaction with IBI. Items are presented on a 1 to 4 Likert scale in which 1 "does not apply to me" and 4 "does apply to me". The total score ranges from 8 to 32. It has adequate psychometric properties, Boß et al. (2016) rate Omega = 0.93 and 0.95 in two different samples.

CONTACTS AND LOCATIONS:
Overall Officials: Azucena García Palacios, Study Chair — Universidad Jaume I; Pedro Vera Albero, Study Director — F.E.D. Psicología Clínica Unitat de Salut Mental Hospital Francesc de Borja; Raquel Escriva Sanchis, Study Chair — F.E.D. Psicología Clínica Unitat de Salut Mental Hospital Francesc de Borja; Clara Bretó García, Study Chair — F.E.D. Psicología Clínica Unitat de Salut Mental Hospital Francesc de Borja
Locations (1):
- Psicología Clínica Unitat de Salut Mental Hospital Francesc de Borja, Tavernes de la Valldigna, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Background] Mira A, Soler C, Alda M, Banos R, Castilla D, Castro A, Garcia-Campayo J, Garcia-Palacios A, Gili M, Hurtado M, Mayoral F, Montero-Marin J, Botella C. Exploring the Relationship Between the Acceptability of an Internet-Based Intervention for Depression in Primary Care and Clinical Outcomes: Secondary Analysis of a Randomized Controlled Trial. Front Psychiatry. 2019 May 10;10:325. doi: 10.3389/fpsyt.2019.00325. eCollection 2019. PMID 31133899
- [Background] Romero-Sanchiz P, Nogueira-Arjona R, Garcia-Ruiz A, Luciano JV, Garcia Campayo J, Gili M, Botella C, Banos R, Castro A, Lopez-Del-Hoyo Y, Perez Ara MA, Modrego-Alarcon M, Mayoral Cleries F. Economic evaluation of a guided and unguided internet-based CBT intervention for major depression: Results from a multi-center, three-armed randomized controlled trial conducted in primary care. PLoS One. 2017 Feb 27;12(2):e0172741. doi: 10.1371/journal.pone.0172741. eCollection 2017. PMID 28241025
- [Background] Montero-Marin J, Araya R, Perez-Yus MC, Mayoral F, Gili M, Botella C, Banos R, Castro A, Romero-Sanchiz P, Lopez-Del-Hoyo Y, Nogueira-Arjona R, Vives M, Riera A, Garcia-Campayo J. An Internet-Based Intervention for Depression in Primary Care in Spain: A Randomized Controlled Trial. J Med Internet Res. 2016 Aug 26;18(8):e231. doi: 10.2196/jmir.5695. PMID 27565118
- [Background] Montero-Marin J, Prado-Abril J, Botella C, Mayoral-Cleries F, Banos R, Herrera-Mercadal P, Romero-Sanchiz P, Gili M, Castro A, Nogueira R, Garcia-Campayo J. Expectations among patients and health professionals regarding Web-based interventions for depression in primary care: a qualitative study. J Med Internet Res. 2015 Mar 10;17(3):e67. doi: 10.2196/jmir.3985. PMID 25757358
- [Background] Karyotaki E, Riper H, Twisk J, Hoogendoorn A, Kleiboer A, Mira A, Mackinnon A, Meyer B, Botella C, Littlewood E, Andersson G, Christensen H, Klein JP, Schroder J, Breton-Lopez J, Scheider J, Griffiths K, Farrer L, Huibers MJ, Phillips R, Gilbody S, Moritz S, Berger T, Pop V, Spek V, Cuijpers P. Efficacy of Self-guided Internet-Based Cognitive Behavioral Therapy in the Treatment of Depressive Symptoms: A Meta-analysis of Individual Participant Data. JAMA Psychiatry. 2017 Apr 1;74(4):351-359. doi: 10.1001/jamapsychiatry.2017.0044. PMID 28241179
- [Background] Mira A, Breton-Lopez J, Garcia-Palacios A, Quero S, Banos RM, Botella C. An Internet-based program for depressive symptoms using human and automated support: a randomized controlled trial. Neuropsychiatr Dis Treat. 2017 Mar 31;13:987-1006. doi: 10.2147/NDT.S130994. eCollection 2017. PMID 28408833
- [Derived] Lorente-Catala R, Font-Furnieles P, Escriva-Sanchis R, Berto-Garcia C, Vera-Albero P, Garcia-Palacios A. Telephone support vs. self-guidance in an Internet-based self-administered psychological program for the treatment of depression: Protocol for a hybrid type 1 effectiveness-implementation randomized controlled trial. Internet Interv. 2024 Apr 20;36:100742. doi: 10.1016/j.invent.2024.100742. eCollection 2024 Jun. PMID 38737981